CLINICAL TRIAL: NCT04438148
Title: Prevalence and Effect of Workplace Stress Among Pediatric Dentists
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Sayed, Principle investigator, Cairo University
Other Study IDs: x643gvu9
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Workplace Stress
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Work-related stress is a pattern of physiological, emotional, cognitive and behavioural reactions to some extremely taxing aspects of work content, work organization and work environment.

Certain work situations are too intense and frequent in nature that exceed an individual's coping capabilities and resources to handle them adequately Dentistry is commonly known as a stressful profession among various occupations. Frequent dealing with different types of patients, working in a very small area for long period of time , exposure to toxic substances , all these factors put the dentist under stress.

Adding to the previous factors, working to uncooperative children with annoying parents, will put pediatric dentistry on the top of the most stressful branches in dentistry.

Stress can affect pedodontists physiologically by increasing their blood pressure, heart rate, breathing rate and excessive sweating which in turn may increase the risk of hypertension and breathing problems.

DETAILED DESCRIPTION:
All Paricipants were informed about the objectives of the study and signed an informed consent before participating in the study.

On the day of work, blood pressure and heart rate will be measured for every pediatric dentist at the beginning of the day before starting any case and will be measured again after 3 hours from continuous work. Then, the two readings will be recorded and compared. This part will help in the physiological assessment of the study.

The psychological part will be assessed by asking the pediatric dentists to answer the questions of the 2 scales. {Appendices (2 &3)}

There will be a specially designed chart for fulfilling the aim of the study designed by the main investigator, this recording chart is formulated to collect the data from the participants.

The recording chart is composed of 3 sections:

The First Section includes sociodemographic data The Second Section includes psychological assessment in which the score gets by each participant is recorded.

The Third Section includes physiological assessment in which the first and second readings of heart rate and blood pressure are recorded and inspected for any change.

ELIGIBILITY:
Inclusion Criteria:

* Both genders are included
* Postgraduate dentists submitting for master and PHD in pediatric dentistry
* Medically free
* The participants who sign the informed consent

Exclusion Criteria:

* Participants taking drugs affecting nervous system
* Fasting participants

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Postgraduate pediatric dentists aged from 25 to 40 years old, medically free
Sampling Method: Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of stress | 6 months
  Cohen percieved stress scale

SECONDARY OUTCOMES:
Degree of stress | 6 months
  Workplace stress scale

OTHER OUTCOMES:
Heart rate | 6 months
  Digital sphygmamanometer
Blood Pressure systolic and diastolic | 6 months
  Digital sphygmamanometer

CONTACTS AND LOCATIONS:
Overall Officials: Maha Sayed, BSc, Principal Investigator — Resident at pediatric dentistry and dental public health department; Shaimaa Sabry, PhD, Study Chair — Lecturer at pediatric dentistry and dental public health department; Walaa Fakher, PhD, Study Chair — Lecturer of Psychiatry, Faculty of Medicine, Cairo University; Randa Youssif, PhD, Study Director — Associate Professer at Pediatric dentistry and dental public health department
Locations (1):
- Cairo University, Cairo, El Manial, Egypt